CLINICAL TRIAL: NCT02469922
Title: Prospective Study Assessing Predictive Value of 18 F-2-fluoro-2-deoxy-D-glucose Fluorodeoxyglucose (FDG) Positron Emission Tomography During Radio-chemotherapy for Locally Advanced Epidermoid Carcinoma of Head and Neck
Brief Title: Positron Emission Tomography (PET) During Radio-chemotherapy to Treat Otorhinolaryngological Cancer
Acronym: TEmPoRAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center Eugene Marquis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-JC-ORLK-TEP; IDRCB : 2013-A01219-36 (Registry Identifier: ANSM)
Record Dates: First submitted 2014-06-25; First posted 2015-06-12 (Estimated); Last update posted 2021-07-27 (Actual); Status verified 2020-07

CONDITIONS: Malignant Neoplasm of Head and Neck; Locally Advanced Malignant Neoplasm
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Positron-Emission Tomography; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Positron emission tomography (Experimental): Two additional PET Scan will be performed at 2 and 4 weeks for the first 30 patients. Then for the other patients only one additional PET-Scan will be performed
  Interventions: Device: Positron emission tomography; Radiation: radiochemotherapy

INTERVENTIONS:
Device: Positron emission tomography
Radiation: radiochemotherapy — Every patients will be treated with radiochemotherapy as a standard of care

SUMMARY:
Open multicentric study assessing predictive value of 18-FDG PET (SUV max) at 20 Gy during radio-chemotherapy, on the loco-regional control after 2 years

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 75 years
* invasive epidermoid carcinoma of head and neck (excluding nasopharyngeal), confirmed by histology
* locally advanced disease (non-metastatic stages AJCC III-IV). AJCC = American Joint Committee on Cancer
* performance status ECOG ≤ 2. ECOG = Eastern Cooperative Oncology Group
* no history of irradiation of the head and neck
* start of radiotherapy within 8 weeks after the pretreatment PET Scan
* no surgery other than biopsy
* pregnancy test: negative for women of childbearing potential
* reliable contraception for a childbearing couple, men and woman must have a reliable contraception during treatment
* signed informed consent form
* patient with national health insurance

Exclusion Criteria:

* prior radiotherapy or chemotherapy
* history of other cancer except: cutaneous non-melanoma tumor and cervix in situ carcinoma
* unstable conditions (cardiovascular, renal, pulmonary) or systemic (lupus erythematosus, scleroderma)
* pregnant patient or patient with breastfeeding
* patient unable to give his consent
* patient under administrative supervision
* patient who participates to another clinical trial on experimental drug
* regular follow-up impossible for various reasons (familial, economical, social, ...)
* diabetes
* accelerated radiotherapy protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2021-01-29 (Actual)

PRIMARY OUTCOMES:
Locoregional relapse | 2 years

SECONDARY OUTCOMES:
Comparison of TEP scan values (Standardized Update Value max, Metabolic Tumor Volume) | pretreatment, 15 days, 29 days, 3 months post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Castelli Joël, Doctor, Principal Investigator — Centre de Lutte Contre le Cancer Centre Eugène Marquis
Locations (5):
- France (5):
  - CHU Brest, Brest
  - Centre jean Bernard - Rue Victor Hugo, Le Mans
  - Hôpital du Scorff, Lorient
  - Centre Eugene Marquis, Rennes
  - Centre d'Oncologie St Vincent - Boulevard de la Boutière, Saint-Grégoire